CLINICAL TRIAL: NCT05552690
Title: Thalassemia Screening by Third Generation Sequencing (TGS): Pilot Study in Thai Population
Brief Title: Thalassemia Screening by Third Generation Sequencing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kuntharee Traisrisilp, Associate Professor, Chiang Mai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 513/2021
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Thalassemia Trait; Thalassemia; Mixed
MeSH Terms: conditions — Thalassemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalassemia screening positive (Other): In this study only 1 group of participants. No comparative. Only description
  Interventions: Procedure: blood draw

INTERVENTIONS:
Procedure: blood draw — 10 ml of blood will be draw to genetic analysis (sequencing)

SUMMARY:
Test globin gene in participants

DETAILED DESCRIPTION:
Recruit individuals who documented as thalassemia carrier or disease and who positive thalassemia screening but unknown mutation.

Blood will be sent for third generation sequencing to review alpha and beta globin gene mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Thalassemia carriers or disease individuals with documented as known globin gene mutation.
2. Thalassemia carriers or disease individuals whose mutation did not retrieve from conventional technique and were assigned as no known mutation

Exclusion Criteria:

-incomplete medical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Validate accuracy of TGS to provide globin gene mutation compared with conventional testing | 6 months after blood test
  Percentage of accuracy to give the mutation diagnosis

SECONDARY OUTCOMES:
Additional mutation added by TGS | 6 months after blood test
  Percentage of mutation are added by sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Maharaj Nakorn ChiangMai Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No